CLINICAL TRIAL: NCT05815537
Title: Development of Functional Spatial Hearing in Reverberation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Father Flanagan's Boys' Home (Other)
Responsible Party: Principal Investigator, Ellen Peng, Research Scientist, Father Flanagan's Boys' Home
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BoysTown
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Spatial Hearing Development

STUDY DESIGN:
Intervention Model Description: There are two arms in the exposure of reverberation for participants. For children (n1=45) and adults (n1=15) assigned to Arm 1, they receive a non-reverberant environment (control) and a low-reverberant environment (intervention A). For children (n2 = 45) and adults (n2 = 15) assigned to Arm 2, they receive the same non-reverberant environment (control) and a high-reverberant environment (intervention B). Both arms of children and adults enrolled perform the same psychoacoustic tasks for outcome assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Reverberation (Experimental): Participants perform psychoacoustic tasks under a low-reverberant environment and a control environment without reverberation.
  Interventions: Other: Low-Reverberation
- High-Reverberation (Experimental): Participants perform psychoacoustic tasks under a high-reverberant environment and a control environment without reverberation.
  Interventions: Other: High-Reverberation

INTERVENTIONS:
Other: Low-Reverberation — The exposure to low-reverberation is by presenting auditory stimuli to participants that are digitally processed to contain auditory cues that sound more or less reverberant, e.g., small classroom.
  Arms: Low-Reverberation
Other: High-Reverberation — The exposure to high-reverberation is by presenting auditory stimuli to participants that are digitally processed to contain auditory cues that sound more or less reverberant, e.g., large lecture hall/auditorium.
  Arms: High-Reverberation

SUMMARY:
The goal of the clinical trial study (Phase 0) is to map out the developmental trajectory of functional spatial hearing abilities in reverberant environments for children with normal hearing between the ages of 6 and 18 years, and to understand the inter-relationships between the three perceptual abilities: auditory object size formation, spatial acuity, and spatial unmasking during typical development. Children are asked to perform psychoacoustic tasks when the auditory stimuli are processed to present in virtual acoustic environments (1) with no reverberation and (2) with one of the two levels of reverberation that emulate everyday indoor environments. The intervention of this clinical study is in the random assignment of one of the two reverberant environments. Researchers will compare these children with a group of normal-hearing adults to anchor matured performances.

ELIGIBILITY:
Inclusion Criteria:

* All individuals within age limits who are typically developing with normal hearing who pass 25 dB HL from 250 Hz to 8000 Hz.

Exclusion Criteria:

* Individuals who fail hearing screen as described above.
* Individuals who have a diagnosed intellectual developmental disability

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Auditory Object Size (Apparent Source Width) | Year 1-3
  Psychoacoustic measure of the smallest detectable change in width of an auditory image in degree angular span in the horizontal plane
Spatial Acuity (Minimum audible angle) | Year 1-3
  Psychoacoustic measure of the smallest detectable angular separation between two auditory objects
Spatial Unmasking (Minimum angular separation) | Year 1-3
  Psychoacoustic measure of the smallest angular separation to gain a target speech benefit in the presence of distracting speech maskers

CONTACTS AND LOCATIONS:
Overall Officials: Z. Ellen Peng, Principal Investigator — Father Flanagan's Boys' Home
Locations (1):
- Boys Town National Research Hospital, Omaha, Nebraska, United States